CLINICAL TRIAL: NCT07258498
Title: Submucosal Injection of Dexamethasone for the Control of Post-operative Sequelae After Mandibular Third Molar Surgery
Brief Title: Submucosal Dexamethasone for Control of Post-operative Pain, Trismus, and Swelling After Mandibular Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PAEC General Hospital, Islamabad (Other)
Responsible Party: Principal Investigator, Kanza Ateeque, Postgraduate Trainee Dr Kanza Ateeque, PAEC General Hospital, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PGHI-IRB (DMe)-RCD-06-068
Record Dates: First submitted 2025-11-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Impacted Mandibular Third Molar Extraction
Keywords: submucosal dexamethasone; impacted mandibular third molar; surgical extraction; pain; swelling; trismus
MeSH Terms: conditions — Pain; Trismus | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Study design: Randomized controlled trial (RCT). Setting: Department of Oral & Maxillofacial Surgery, Pakistan Atomic Energy Commission General Hospital, Islamabad.
  Duration: 12 months (after approval of synopsis from CPSP)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): submucosal injection of dexamethasone would be used in this study to prevent post-operative pain , swelling and trismus in patient having surgical extraction of impacted mandibular third molars.
  Interventions: Drug: Dexamethasone
- Normal saline (placebo) (Placebo Comparator): Out of 70 patients 35 patients would be given submucosal injection of normal saline as a placebo.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexamethasone — In this study submucosal injection of dexamethasone would be given to the patient 30 minutes before surgical extraction of impacted mandibular third molar surgery to reduce pain, swelling and trismus, thus to minimize patient's discomfort after surgery, so that the patients could pursue their daily activities without delay
  Arms: Dexamethasone
Drug: Normal Saline — submucosal injection of normal saline (N/S) would not reduce trismus, swelling, and pain
  Arms: Normal saline (placebo)

SUMMARY:
Purpose: The aim of this study is to determine the efficacy of submucosal injection of dexamethasone in reducing pain, swelling and trismus, thus to minimize patient's discomfort after surgery, so that the patients could pursue their daily activities without delay. Moreover, the submucosal injection is convenient to the patient and surgeon both, as it is injected after application of local anesthesia and easily administered. OBJECTIVES: To evaluate the outcome of submucosal injection of 4mg/ml dexamethasone in comparison with submucosal injection of normal saline (N/S) on mean post-operative pain, trismus and swelling following mandibular third molar surgery.

DETAILED DESCRIPTION:
OPERATIONAL DEFINITIONS:

Pain: Post-operative pain outcome when measured using Visual Analogue Scale (VAS) would determine the subjective pain experience of patients. VAS is a straight, 10 cm long horizontal line. VAS represents continuous pain intensity, where the left end of the line indicates "no pain," while the right end denotes "worst pain imaginable." Patients indicate their level of pain (in cm) by marking a single point on the line.

Swelling: Post-operative facial swelling would be assessed by using Gabka and Matsumara technique. Linear distance between angle of the mandible to lateral corner of the eye (A), distance between tragus to corner of the mouth (B), and distance between tragus to soft tissue pogonion (C) would be quantified in millimeters using measuring tape. The sum of these measurements would be calculated as facial dimension and used to measure the level of swelling in millimeters.

Trismus: Trismus i.e., reduced mouth opening would be quantified in millimeters by measuring interincisal distance at maximum mouth opening using a vernier caliper. Normal mouth opening ranges from 40 to 60 mm. Mouth opening less than 40 mm is considered trismus.

HYPOTHESIS:

Submucosal injection of 4mg/ml dexamethasone will result in lower mean postoperative pain, reduced trismus and less swelling after mandibular third molar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cases of impacted mandibular third molar according to Pell and Gregory classification (class l, 2. 3 and A. B, C)
* Both genders (male and female)
* Age limit: 18 - 45 years

Exclusion Criteria:

* Patients with pericoronitis.
* Patients with known allergy to corticosteroids.
* Medically compromised patients.
* Current pregnancy.
* Lactating women.
* Use of medication by the patients that could interfere with the healing process.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
measurement of post-operative pain, in patients who have undergone surgery for impacted mandibular third molars. | from enrolment to 7th post operative day
  Pain: Post-operative pain outcome when measured using Visual Analogue Scale (VAS) would determine the subjective pain experience of patients. VAS is a straight, 10 cm long horizontal line. VAS represents continuous pain intensity, where the left end of the line indicates "no pain," while the right end denotes "worst pain imaginable." Patients indicate their level of pain (in cm). by marking a single point on the line.
measurement of post-operative trismus in patients who have undergone surgery for impacted mandibular third molars. | From enrollment to the 7th Postoperative day
  Trismus i.e., reduced mouth opening would be quantified in millimeters by measuring interincisal distance at maximum mouth opening using a vernier caliper. Normal mouth opening ranges from 40 to 60 mm. Mouth opening less than 40 mm is considered trismus.
measurement of post-operative swelling in patients who have undergone surgery for impacted mandibular third molars. | from enrolment to 7th post operative day
  Swelling: Post-operative facial swelling would be assessed by using Gabka and Matsumara technique. Linear distance between angle of the mandible to lateral corner of the eye (A), distance between tragus to corner of the mouth (B), and distance between tragus to soft tissue pogonion (C) would be quantified in millimeters using measuring tape. The sum of these measurements would be calculated as facial dimension and used to measure the level of swelling in millimeters.

SECONDARY OUTCOMES:
demographic data (name, age, gender) | from enrolment to 7th post operative day
  name, age, gender would be used to assess the effects of demographic data on post operative sequelae
tooth number of impacted tooth according to FDI tooth numbering system, type of impaction | from enrolment to 7th post operative day
  tooth number of impacted tooth according to FDI tooth numbering system, type of impaction according to pell and gregory classification would be used to assess any effect of these outcomes on post-operative sequelae after mandibular third molar surgery.
No. of Paracetamol 500 mg tablets taken orally postoperatively | from enrolment to 7th post operative day
  No. of Paracetamol 500 mg tablets taken orally postoperatively would be used to assess if patient was pain free or had pain post-operatively following impacted mandibular third molar surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kanza Ateeque, BDS, Principal Investigator — PAEC General Hospital, Islamabad
Locations (1):
- PAEC General Hospital, Islamabad, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No
As the hospital where this study is being conducted does allow to share any collected data with other researchers due to patient confidentiality